CLINICAL TRIAL: NCT05663463
Title: Seasonal Influenza Vaccine High Dose Boosting in Solid Organ Transplant Recipients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: NA-Influenza
Record Dates: First submitted 2022-12-12; First posted 2022-12-23 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Solid Organ Transplant
MeSH Terms: interventions — Influenza Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- booster group (Experimental): Participants who have undergone a solid organ transplant will receive two doses of an inactivated high dose influenza vaccine
  Interventions: Drug: Fluzone High-Dose - 2 doses
- Control group (Active Comparator): Participants who have undergone a solid organ transplant will receive one dose of inactivated high dose influenza vaccine followed by a placebo injection
  Interventions: Drug: Fluzone High-Dose - 1 dose of HD

INTERVENTIONS:
Drug: Fluzone High-Dose - 2 doses — 2 doses of the High-Dose (HD) influenza vaccine separated by 4-6 weeks For 2023-2024 influenza season the influenza quadrivalent HD vaccine was used. For 2024 -2025 influenza season the influenza trivalent HD vaccine will be used.
  Arms: booster group
Drug: Fluzone High-Dose - 1 dose of HD — 1 dose of the High Dose (HD) influenza vaccine, followed by a placebo injection 4-6 weeks later For 2023-2024 influenza season the influenza quadrivalent HD vaccine was used. For 2024 -2025 influenza season the influenza trivalent HD vaccine will be used.
  Arms: Control group

SUMMARY:
In solid organ transplant (SOT) the receipt of influenza vaccine in an influenza season is associated with decreased disease severity as demonstrated by the presence of pneumonia and ICU admissions. Different strategies have been assessed to optimize vaccine efficacy and immunogenicity of the influenza vaccine in the solid organ transplant recipient (SOTR). The primary objective of the study is to evaluate the immunogenicity of 2 doses of the high dose influenza vaccine utilizing neutralizing antibody assays. A control group receiving 1 HD influenza vaccine will be included.

ELIGIBILITY:
Inclusion Criteria:

* >=18 years old who underwent a solid organ transplant (Liver, lung, heart, kidney, pancreas) > 1 year prior to enrollment
* At least 1-year post-transplant
* Able and willing to provide informed consent
* Able and willing to undergo all study activities throughout the duration of the study

Exclusion Criteria:

* Confirmed pregnancy
* Receipt of ATG or carfilzomib within the past 3 months
* Receipt of rituximab within the past 3 months
* Receipt of basiliximab within the past 3 months
* Prednisone dose >= 20 mg/day at the time of enrollment
* History of a severe allergy to influenza vaccine (i.e. Guillain Barre syndrome, anaphylaxis or angioedema)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2023-09-11 (Actual); Primary Completion 2025-06-16 (Actual); Study Completion 2025-06-16 (Actual)

PRIMARY OUTCOMES:
Neutralizing antibody levels- Immunogenicity | Baseline
  Geometric mean titers and geometric mean fold rise from baseline of homologue neutralizing antibodies in reporter microneutralization will be measured and compared across groups.
Neutralizing antibody levels- Immunogenicity | 4-6 weeks after dose 1
  Geometric mean titers and geometric mean fold rise from baseline of homologue neutralizing antibodies in reporter microneutralization will be measured and compared across groups.
Neutralizing antibody levels- Immunogenicity | 3 months after 2nd dose
  Geometric mean titers and geometric mean fold rise from baseline of homologue neutralizing antibodies in reporter microneutralization will be measured and compared across groups.

SECONDARY OUTCOMES:
clinical outcome- pneumonia | 2 years
  assess clinical outcome associated with an influenza infection such as pneumonia rates during the 2023-2024 and 2024-2025 influenza seasons.
clinical outcome- hospitalization rates | 2 years
  assess clinical outcome associated with an influenza infection such as hospitalization rates during the 2023-2024 and 2024-2025 influenza seasons.
clinical outcome- ICU admissions | 2 years
  assess clinical outcome associated with an influenza infection such as ICU admission rates during the 2023-2024 and 2024-2025 influenza seasons.
clinical - death rates | 2 years
  assess clinical outcome associated with an influenza infection such as death rates during the 2023-2024 and 2024-2025 influenza seasons.

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Fontana, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States